CLINICAL TRIAL: NCT06539052
Title: A Model to Improve the Screening and Linkage to Care of HDV Infection in Migrant Living in Southern Italy Taking Advantage of HDV Reflex Testing: MIGrant Reflex Test HDV (MIGRED) Project
Brief Title: MIGrant Reflex Test HDV (MIGRED) Project
Status: Not yet recruiting | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Nicola Coppola, Chief of Infectoius Diseases Unit, University of Campania Luigi Vanvitelli
Other Study IDs: MIGRED
Record Dates: First submitted 2024-07-23; First posted 2024-08-06 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Hepatitis D Virus Infection
MeSH Terms: conditions — Hepatitis D

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- migrants: All migrants, documents or undocumented migrants, and low-income refugees belonging to the infectious disease centers of the university centers participating in the project will be enrolled.
  All HBsAg-positive subjects will be linked to the tertiary centers. The cultural mediator will accompany the migrants testing positive to the screening to stage the liver disease and to start the therapeutic management of subjects with HBV infection and HBV HDV co-infection according to international guidelines.
  In the Retrospective phase of the project about 2000 stored samples of migrant enrolled in a previous study will be re-tested for HBsAG, HCV Ab and HIV ab. In the same blood sample testing positive for HBsAg, anti-HDV will be tested; in cases of anti-HDV positivity the same serum sample will be collected to test HDV RNA.
  Interventions: Diagnostic Test: anti-HDV positive with the reflex testing methodology

INTERVENTIONS:
Diagnostic Test: anti-HDV positive with the reflex testing methodology — Rate of screening for HBsAg in all migrants attending to one of the center participating to the project rate of screening for anti-Delta in all HBsAg patients identified rate of anti-Delta-positivity in HBsAg-positive subjects rate of linkage-to-care at one of the infectious disease center participating to the project rate of HDV-RNA testing in all anti-Delta positive subjects rate of treatment for HDV in all HDV-RNA-positive subjects Rate of screening for HIV Ab in all migrants attending to one of the center participating to the project Rate of screening for HCV Ab in all migrants attending to one of the center participating to the project.

SUMMARY:
Our research team has executed a robust strategy to improve viral hepatitis detection and linkage to care in migrants, contributing to the improvement of knowledge on the clinical and virological future of viral hepatitis in this population difficult to reach and manage. Our hypothesis is that the extension of our model to three other large university clinical centers operating in southern Italy and the use of HDV reflex testing for HBsAg-positive subjects will allow the implementation of knowledge on prevalence of HDV in migrants living in southern Italy and coming from HDV endemic areas. Precisely, the investigators will involve the Department of Infectious Diseases of the University of Bari, that of the University of Catanzaro and that of the University of Palermo with expertise in the management of infectious diseases in the migratory context and with whom the investigators have previously collaborated in other areas.

It is expected to enroll at least 7500 patients. The project will last 18 months.

Diagnosis and treatment of HDV infection in migrants will reduce the circulation of HDV in low endemic regions such as our region. Follow-up of HDV-infected individuals and reducing the rate of new infections among migrants will reduce the number of people who will experience complications related to HDV infection, such as decompensated liver cirrhosis and carcinoma hepatocellular. All this will determine benefits for the Italian public health system.

DETAILED DESCRIPTION:
Hepatitis D virus (HDV) infection, which occurs only in subjects with hepatitis B infection, increases the risk of hepatocellular carcinoma (HCC), decompensated cirrhosis, and mortality compared to hepatitis B virus (HBV) mono-infection. Therefore, estimates the prevalence of HDV infection and disease burden are essential to investigate models to find coinfected individuals more effectively and in an efficient way. Diagnosis of HDV allows to reduce the risk of disease progression and prevent HDV transmission, allows to intervene with antiviral treatment and allows to follow-up HDV positive subjects with ultrasound for HCC surveillance [1-4]. The data on the prevalence of HDV worldwide is unclear, with an estimated prevalence of anti-Delta-positivity in HBsAg positive patients of 4.5%-13% and an estimated number of anti-Delta-subjects of 8,2-60 million [5-6]. These variable estimates may be due in part to the fact that not all HBsAg-positive subjects were screened for anti-Delta. All the strategies for the improvement of the rate of screening of HBsAg-positive-subjects may improve the knowledge on the prevalence of HDV worldwide, especially in the high endemic populations. Recently, one of the strategies that has shown good results in the identification of HDV infection is the use of anti HDV reflex testing [4]. However, HDV is highly endemic in several African countries and in some countries in South America, the Middle East, central and northern Asia, and Eastern Europe [7]. A systematic review of the prevalence of HDV infection in HBsAgpositive populations in sub Saharan Africa showed a pooled seroprevalence in HBsAg-positive general populations and in patients with liver disease of 7.33% and 9.57%, respectively in western Africa, of 25.6% and 37.8% in central Africa, and of 0.05% in the general populations of eastern and southern Africa [8]. In Italy the prevalence of HDV infection in HBsAg-positive subjects ranges from 9.7 to 12%, with evidence of an increasing prevalence of HDV infection in the immigrant population in recent years [9-15]. Probably, this happened because for its geographical position in the center of the Mediterranean Sea, Italy has been greatly involved in immigration from Africa, in particular from sub-Saharan Africa, and also from Asia and Eastern Europe; for example from January 2023 until September 2023 in Italy are arrived about 128,000 migrants and most of them coming from Sub-Saharan Africa and East Europe, prevalence (Situation Mediterranean Situation (unhcr.org), all areas with high HDV prevalence, The majority of these migrants arrived, as first site, in Southern Italy, Sicily, Apulia, Calabria and Campania. However, few data have been published so far on the prevalence of HDV infection in immigrant populations in Western countries and in Italy and even poorer is the information on the virological and clinical aspects of HDV infection in this population.

Our research group performed a valid strategy to improve the detection for viral hepatitis and the link to care in migrants, contributing to the improvement of knowledge on clinical and virological futures of viral hepatitis in this population difficult to reach and to manage [1-3]. Our hypothesis is that the extension of our model in other three large university clinical centers operating in southern Italy and the use of the HDV reflex testing for HBsAg-positive individuals will allow to implement the knowledge on the HDV prevalence in migrants living in southern Italy and coming from endemic areas for HDV. Precisely, the investigators will involve the Department of Infectious Diseases of the University of Bari, that of the University of Catanzaro and that of the University of Palermo with expertise in the management of infectious diseases in migrant and with which the investigators previously collaborated in other setting.The investigators performed a retrospective and prospective multicenter project lasting 18 months involving the 4 largest University clinical Centers for Infectious Diseases (ID) in southern Italy:

Departments of ID of the University of Napoli L.Vanvitelli (project coordinator), of the University of Bari, of the University of Catanzaro and of the University Palermo.

At this time they are not involved in any other projects involving screening and linkage to care of HDV infection.

Each of these tertiary center is associated to 1st level clinical centers, that are centers of general practice clinics attended mainly by migrants for low back pain, headache, itching, cough, hypertension and allergy symptoms. These first-level centers are linked with the Italian humanitarian organizations which welcome needy migrants. The organization of these clinics involves the presence of a physhycian expert in the management of infectious diseases in migrants, a nurse and a cultural mediator. This last figure is fundamental in explaining the epidemiological, clinical and collective health reasons that make it necessary to screen for hepatitis viruses which are endemic in their areas of origin.

Screening process All sample of migrants relating to the infectious diseases clinic of the centers participating in the project will be collected.

To improve the rate of enrollment, the physicians, with the help of cultural mediators, will explain to the what are the main sexually and parenterally transmitted infectious diseases endemic in their countries of origin and will be information on the routes of transmission of theses. The information/education will be done through brochures with pictures and explanations translated into English, French and Swahili. The migrants, who agreed to join the project, signed an informed consent written in the immigrant's own language and filled out an anonymous questionnaire administered by the research investigators with the assistance of a cultural mediator on the demographic data, date of immigration, socioeconomic status (level of education), religion, cohabitation details, sexual orientation and practices including condom use, history of HBV vaccination, surgery, dental care, tattooing, body piercing, use of drugs, blood transfusion, tribal rituals, abortion and information on previously documented personal and family infections of HBV, HDV, HCV and HIV. The data relating to the epidemiological characteristics will collected in an electronic database.

A blood sample will be collected. The cultural mediator will support the clinicians and the nurses who will collect the blood sample to ensure that the migrant fully and freely understands the reasons of the screening.

An epidemiological data sheet will be associated with the blood sample. Every center will carry out HBsAg testing on the blood samples collected. The HBsAg positivity will be the trigger to start the HDV reflex testing cascade: in the same blood sample testing positive for HBsAg, anti-HDV will be tested; in cases of anti-HDV positivity the same serum sample will be collected to test HDV RNA.

HDV RNA will be performed at the molecular biology laboratory of the Department of ID of the University of Naples (project coordinator) according to standard methods. Once a month, the samples tested anti-HDV positive with the reflex testing methodology will be carried on dry ice at a controlled temperature to the reference center for the virological tests. For subjects with positive HDV viremia the investigators will proceed for HDV genotyping on the same serum sample.

The same sample will also be tested for HIV and HCV, any positivity will be communicated to the reference.

All HBsAg-positive subjects will be linked to the tertiary centers. The cultural mediator will accompany the migrants testing positive to the screening to stage the liver disease and to start the therapeutic management of subjects with HBV infection and HBV HDV co-infection according to international guidelines.

In the Retrospective phase of the project about 2000 stored samples of migrant enrolled in a previous study will be re-tested for HBsAG, HCV Ab and HIV ab. In the same blood sample testing positive for HBsAg, anti-HDV will be tested; in cases of anti-HDV positivity the same serum sample will be collected to test HDV RNA.

In the regions of southern Italy where the project will take place, that is Campania, Apulia, Calabria and Sicily, approximately 128,000 migrants arrived from January 2023 until September 2023 (https://data2.unhcr.org/en/situations/mediterranean). In consideration of the economic availability of the project the investigators aim to evaluate approximately 7,500 migrants. the investigators hypothesize to enroll 7500 migrants. Of these 7500, the investigators hypothesize that about 4500 have already been screened for HBsAg, HCV Ab, HIV Ab, while 3000 must been screened for these viruses. The project will last 18 months and for all 7500 enrolled migrants will be carried out HBsAg, HIV Ab and HCV Ab screening. Samples positive for HBsAg will be tested for HDV at the same time as the positive result of HBsAg. Considering a prevalence of HBsAg-positivity of 10% in migrant population, the investigators hypothesize to identify 750 HBsAg-positive subjects. Considering that the prevalence of HDV in HBsAg positive subjects in Africa is estimated of approximately 9%, the investigators hypothesize to identify 68 anti-HDV positive subjects.

ELIGIBILITY:
Inclusion Criteria:

* All migrants, documents or undocumented migrants, and low-income refugees belonging to the infectious disease centers of the university centers participating in the project will be enrolled. aged > 18 years subjects who have given informed consent to carry out blood sampling and for the collection of epidemiological data

Exclusion Criteria:

* all migrants < 18 years of age who have not given informed consent for the collection of the blood sample and/or epidemiological data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HDV reflex testing is already performed in specific regions (Spain, France, Brazil, Sweden, Canada), but not at the national level. There are few data on the applicability of this methodology in migrants coming from HDV endemic areas therefore we think that testing this model in this population is useful. The diagnosis and treatment of HDV infection in migrants will reduce the circulation of HDV in low endemic regions such as our region. The follow up of subjects with HDV infection and the reduction in the rate of new infections among migrants, will reduce the number of people who will present complications related to HDV infection, such as decompensated liver cirrhosis and hepatocellular carcinoma. All this will determine benefits to the Italian public health system.
Sampling Method: Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Number of anti-Delta-positive subjects connected to tertiary services. | 1 month
  Clinical recording of referrals and confirmation of successful connection through digital medical records
Detection rate of HDV RNA. | 1 month
  quantitative Test RT-PCR (Reverse Transcription Polymerase Chain Reaction).
Number of subjects evaluated for therapy. | 1 month
  Clinical patient records and standardized medical assessments
Prevalence of anti-Delta positivity in different demographic categories. | 1 month
  Demographic questionnaires
Distribution of clinical (e.g., ALT/AST levels, liver fibrosis) features based on anti-Delta positivity. | 1 month
  Measuring instrument: Standardized laboratory tests (blood tests, virological tests) and diagnostic tools (ultrasounds, fibroscans).
Assessment of virological (e.g., HBV viral load) features | 1 month
  This outcome measure will assess HBV viral load in anti-Delta positive subjects and how it varies with HDV-RNA positivity. HBV viral load will be quantified using specific and standardized virological tests.
  Measurement tool: Laboratory testing for HBV viral load, such as polymerase chain reaction (PCR) quantification.
  Data aggregation: Viral load data will be aggregated and presented as mean viral load, median, and distribution of viral loads in HDV-RNA positive subjects. Descriptive statistics will include minimum, maximum, means, and standard deviations
Number of HBsAg positive subjects who are also HIV Ab positive and/or HCV Ab positive. | 1 month
  Enzyme-Linked Immunosorbent Assay (ELISA) test for HIV Ab and HCV Ab.
Distribution of demographic characteristics (age, sex, geographical origin) | 1 month
  This measure will assess how demographic characteristics (age, sex, geographic origin) are distributed among anti-Delta positive subjects based on HDV-RNA positivity.
  * Measurement tool: Demographic questionnaires completed by participants.
  * Data aggregation: Data will be aggregated by age, gender, and geographic origin, and presented in frequency tables and descriptive statistics.
Distribution of Virological Features | 1 month
  This measure will assess how virological features (e.g., HBV and HDV viral load) are distributed among anti-Delta positive subjects based on HDV-RNA positivity.
  * Measurement tool: Laboratory testing for HDV-RNA using RT-PCR (Reverse Transcription Polymerase Chain Reaction) and virological tests for HBV viral load.
  * Data Aggregation: Data will be aggregated by viral load and presented in frequency tables and descriptive statistics.
Distribution of clinical features | 1 month
  This measure will assess how clinical features (e.g., ALT/AST levels, liver fibrosis) are distributed among anti-Delta positive subjects based on HDV-RNA positivity.
  * Measurement Tool: Standardized clinical examinations, including blood tests for ALT/AST levels and liver fibrosis assessments via fibroscan.
  * Data aggregation: Data will be aggregated for each clinical parameter and presented in frequency tables and descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Coppola, MD, Principal Investigator — Università della Campania Luigi Vanvitelli

IPD SHARING:
Plan to Share IPD: Undecided
data will be disseminated only in a strictly anonymous and aggregated form at scientific conferences or through scientific or statistical publications. They may be shared with other centers in the context of scientific discussions or in national and international consortia to draw up revisions of the current guidelines..data may be transferred to third countries outside the European Union subject to subjects consent. The transfer of data will take place in compliance with the rules set out in Chapter V of the GDPR EU 2016/679 (art. 44 et seq.), in such a way as to guarantee an adequate level of protection of personal data established in the contractual phase, also through specific clauses

REFERENCES:
- [Result] Beguelin C, Moradpour D, Sahli R, Suter-Riniker F, Luthi A, Cavassini M, Gunthard HF, Battegay M, Bernasconi E, Schmid P, Calmy A, Braun DL, Furrer H, Rauch A, Wandeler G; Swiss HIV Cohort Study. Hepatitis delta-associated mortality in HIV/HBV-coinfected patients. J Hepatol. 2017 Feb;66(2):297-303. doi: 10.1016/j.jhep.2016.10.007. Epub 2016 Oct 14. PMID 27746337
- [Result] Roulot D, Brichler S, Layese R, BenAbdesselam Z, Zoulim F, Thibault V, Scholtes C, Roche B, Castelnau C, Poynard T, Chazouilleres O, Ganne N, Fontaine H, Gournay J, Guyader D, Le Gal F, Nahon P, Roudot-Thoraval F, Gordien E; Deltavir study group. Origin, HDV genotype and persistent viremia determine outcome and treatment response in patients with chronic hepatitis delta. J Hepatol. 2020 Nov;73(5):1046-1062. doi: 10.1016/j.jhep.2020.06.038. Epub 2020 Jul 4. PMID 32634548
- [Result] Fattovich G, Giustina G, Christensen E, Pantalena M, Zagni I, Realdi G, Schalm SW. Influence of hepatitis delta virus infection on morbidity and mortality in compensated cirrhosis type B. The European Concerted Action on Viral Hepatitis (Eurohep). Gut. 2000 Mar;46(3):420-6. doi: 10.1136/gut.46.3.420. PMID 10673308
- [Result] Romeo R, Del Ninno E, Rumi M, Russo A, Sangiovanni A, de Franchis R, Ronchi G, Colombo M. A 28-year study of the course of hepatitis Delta infection: a risk factor for cirrhosis and hepatocellular carcinoma. Gastroenterology. 2009 May;136(5):1629-38. doi: 10.1053/j.gastro.2009.01.052. Epub 2009 Jan 29. PMID 19208358
- [Result] Stockdale AJ, Kreuels B, Henrion MYR, Giorgi E, Kyomuhangi I, de Martel C, Hutin Y, Geretti AM. The global prevalence of hepatitis D virus infection: Systematic review and meta-analysis. J Hepatol. 2020 Sep;73(3):523-532. doi: 10.1016/j.jhep.2020.04.008. Epub 2020 Apr 23. PMID 32335166
- [Result] Miao Z, Zhang S, Ou X, Li S, Ma Z, Wang W, Peppelenbosch MP, Liu J, Pan Q. Estimating the Global Prevalence, Disease Progression, and Clinical Outcome of Hepatitis Delta Virus Infection. J Infect Dis. 2020 Apr 27;221(10):1677-1687. doi: 10.1093/infdis/jiz633. PMID 31778167
- [Result] Rizzetto M, Ponzetto A, Forzani I. Hepatitis delta virus as a global health problem. Vaccine. 1990 Mar;8 Suppl:S10-4; discussion S21-3. doi: 10.1016/0264-410x(90)90207-3. PMID 2183511
- [Result] Stockdale AJ, Chaponda M, Beloukas A, Phillips RO, Matthews PC, Papadimitropoulos A, King S, Bonnett L, Geretti AM. Prevalence of hepatitis D virus infection in sub-Saharan Africa: a systematic review and meta-analysis. Lancet Glob Health. 2017 Oct;5(10):e992-e1003. doi: 10.1016/S2214-109X(17)30298-X. PMID 28911765
- [Result] Sagnelli E, Stroffolini T, Mele A, Imparato M, Sagnelli C, Coppola N, Almasio PL. Impact of comorbidities on the severity of chronic hepatitis B at presentation. World J Gastroenterol. 2012 Apr 14;18(14):1616-21. doi: 10.3748/wjg.v18.i14.1616. PMID 22529690
- [Result] Sagnelli E, Sagnelli C, Pisaturo M, Macera M, Coppola N. Epidemiology of acute and chronic hepatitis B and delta over the last 5 decades in Italy. World J Gastroenterol. 2014 Jun 28;20(24):7635-43. doi: 10.3748/wjg.v20.i24.7635. PMID 24976701
- [Result] Stroffolini T, Sagnelli E, Sagnelli C, Russello M, De Luca M, Rosina F, Cacopardo B, Brancaccio G, Furlan C, Gaeta GB, Licata A, Almasio PL; behalf of EPACRON study group. Hepatitis delta infection in Italian patients: towards the end of the story? Infection. 2017 Jun;45(3):277-281. doi: 10.1007/s15010-016-0956-1. Epub 2016 Nov 5. PMID 27817147
- [Result] Gaeta GB, Stroffolini T, Smedile A, Niro G, Mele A. Hepatitis delta in Europe: vanishing or refreshing? Hepatology. 2007 Oct;46(4):1312-3. doi: 10.1002/hep.21816. No abstract available. PMID 17894318
- [Result] Sagnelli E, Stroffolini T, Mele A, Imparato M, Almasio PL; Italian Hospitals' Collaborating Group. Chronic hepatitis B in Italy: new features of an old disease--approaching the universal prevalence of hepatitis B e antigen-negative cases and the eradication of hepatitis D infection. Clin Infect Dis. 2008 Jan 1;46(1):110-3. doi: 10.1086/524074. PMID 18171224
- [Result] Sagnelli C, Sagnelli E, Russo A, Pisaturo M, Occhiello L, Coppola N. HBV/HDV Co-Infection: Epidemiological and Clinical Changes, Recent Knowledge and Future Challenges. Life (Basel). 2021 Feb 22;11(2):169. doi: 10.3390/life11020169. PMID 33671730
- [Result] Coppola N, Alessio L, Onorato L, Sagnelli C, Sagnelli E, Pisaturo M. HDV infection in immigrant populations. J Med Virol. 2019 Dec;91(12):2049-2058. doi: 10.1002/jmv.25570. Epub 2019 Aug 27. PMID 31429940